CLINICAL TRIAL: NCT07304531
Title: First To Know Pregnancy Test Clinical Evaluation Protocol
Brief Title: First To Know Pregnancy Test - Clinical Evaluation Protocol
Status: Recruiting | Type: Observational
Sponsor: NOWDiagnostics, Inc. (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-STDY-8001-01
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Detection
Keywords: NOWDx First To Know Pregnancy Detection Test
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Cohort A1 - Pre-menopausal women ages 14-40: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, ages 14-40
  Interventions: Device: Diagnostic Test
- Cohort A2 - Peri-menopausal women ages 41-55: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, ages 41-55
  Interventions: Device: Diagnostic Test
- Cohort A3 - Post-menopausal women ages >55: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, age over 55
  Interventions: Device: Diagnostic Test
- Cohort B1 - Subset of Cohort A1 Pre-menopausal women ages 14-40: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, ages 14-40
  Interventions: Device: Diagnostic Test
- Cohort B1 - Subset of Cohort A2 - Peri-menopausal women ages 41-55: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, ages 41-55
  Interventions: Device: Diagnostic Test
- Cohort B3 - Subset of Cohort A3 - Post-menopausal women ages >55: Participants must be a mixture of English and Spanish speaking, geographically diverse, ethnically and racially diverse, economically diverse, and with different levels of educations, age over 55
  Interventions: Device: Diagnostic Test

INTERVENTIONS:
Device: Diagnostic Test — For this observational trial , the Intervention of interest is the First To Know Pregnancy Test

SUMMARY:
This study is evaluating the ADEXUSDx® hCG CLIA moderately complex, FDA-cleared test for potential over the counter (OTC) use and marketing as the First To Know® (FTK) Pregnancy test. The investigational FTK Pregnancy test will be used to assess its clinical performance in the intended use population (i.e., lay users) through self-testing in a simulated home setting.

DETAILED DESCRIPTION:
The Investigational First to Know® Pregnancy test has been adapted from the CLIA moderately complex, FDA-cleared ADEXUSDx® hCG test for clinical evaluation to enable lay users to self-test in a simulated home environment in the US. The First To Know® Pregnancy test is currently CE marked in the EU for OTC use. The assays remain identical in their formulation and performance characteristics.

The clinical evaluation includes lay users self-testing and additional blood being drawn for comparator testing. All negative test results will be followed up for outcome. All subjects with positive test results or reporting negative results later resulted in pregnancy will be confirmed by obtaining data from standard of care assessment(s) for diagnosis of pregnancy.

Two (2) cohorts are planned to assess:

Cohort A: Cross sectional cohort evaluating clinical performance with enrollment up to 100 pregnant subjects across three (3) age groups conducted at clinical sites. Tests will be read and interpreted by the lay user. Blood will be collected at the time of testing for comparator method testing. Positive test results will be confirmed by obtaining data from standard of care assessment(s) for diagnosis of pregnancy.

Cohort A1: pre-menopausal women age 14-40

Cohort A2: peri-menopausal women age 41-55

Cohort A3: post-menopausal women age >55

Cohort B: Duplicate testing cohort designed to evaluate accuracy and precision in lay users. A subset of a minimum of 100 participants from Cohort A will co-enroll into Cohort B and conduct duplicate testing using the First To Know® Pregnancy test. Participants will independently self-administer two tests consecutively and visually interpret the results without assistance.

Enrollment will reflect the observed prevalence of positive and negative pregnancy results in Cohort A, ensuring adequate representation across all age cohorts (pre-menopausal, peri-menopausal, and post-menopausal). The results from the first test will be used to assess accuracy, while the second test will evaluate precision and agreement with the first test.

ELIGIBILITY:
Inclusion Criteria:

* Females whose pregnancy status is unknown (e.g., have not used urine test at home)
* Age Selection - must meet one of the following age groups:
* Cohort A1 - Pre-menopausal: ≥14 years of age and ≤ 40 years of age with menstrual cycles (cycle lengths of 25-35 days)
* Cohort A2 - Peri-menopausal: ≥41 years of age and ≤ 54 years of age
* Cohort A3 - Post-menopausal: ≥55 years of age
* Not menstruating at the time of the initial study visit
* Must be willing to complete all study activities, provide all specimens/samples, and conduct all required testing
* Willing to provide information regarding the diagnosis of pregnancy or details from their standard of care follow-up visit after initial visit
* Sexually active
* Not using contraceptives
* English/Spanish speaking

Exclusion Criteria:

* Males
* Females <14 years of age
* Recent pregnancy within the past 6 months
* Trophoblastic disease or non-trophoblastic neoplasms
* Downs syndrome (trisomy 21)
* People with limited or no reading skills
* Amenorrhea not related to peri or post menopause
* Use of medications or hormonal contraceptives that may interfere with hCG levels at the time of testing (e.g., Gonadotropins: Luteinizing hormone)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender females
Study Population: Female residents of the United States who elect to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1705 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy and sensitivity of the First To Know Pregnancy test compared to a legally marketed quantitative blood-based hCG assay | Through study completion, an average of 6 months
  Evaluate the accuracy and sensitivity of the First To Know Pregnancy test compared to a legally marketed quantitative blood-based hCG assay (e.g., Siemens Dimension® hCG Flex® Reagent Cartridge, Roche Cobas® Elecsys HCG STAT) as the clinical comparator

SECONDARY OUTCOMES:
Assess the performance of the FTK Pregnancy test near the cutoff range | Through study completion, an average of six months
  Calculate the sensitivity and specificity of the First To Know Pregnancy test near the cutoff range.
Evaluate the test's specificity in pre-menopausal, peri-menopausal and post-menopausal women | through study completion, an average of 6 months
  Evaluate the test's specificity in pre-menopausal, peri-menopausal and post-menopausal women to assess false positives
Follow subjects to confirm pregnancy status | through study completion, an average of 6 months
  Follow subjects to confirm pregnancy status to compute accuracy of the First To Know Pregnancy Test.
Evaluate lay user performance under real-world conditions | through study completion, an average of 6 months
  Calculate invalid rate for lay users performing the First To Know Pregnancy test under real world conditions.
Assess the usability of the test | through study completion, an average of 6 months
  Calculate useability statistics for lay users performing the First To Know Pregnancy test under real world conditions through their First To Know Pregnancy Useability Questionnaire Responses
Evaluate testing precision | through study completion, an average of 6 months
  Compute concordance in duplicate tests performed by a subset of subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Matrix Clinical Research Los Angeles, Los Angeles, California
  - ERA Health Research, Midland, Texas

IPD SHARING:
Plan to Share IPD: No